CLINICAL TRIAL: NCT06636123
Title: GZ17-6.02 in Advanced Castration-Resistant Prostate Cancer (CRPC) After Progression on Anti-Androgen Therapy
Brief Title: GZ17-6.02 in Advanced CRPC After Progression on Anti-Androgen Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23-20417; HM20030070 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Investigational Agent Administration (Experimental): GZ17-6.02: 375mg twice daily
  Interventions: Drug: Investigational Agent Administration

INTERVENTIONS:
Drug: Investigational Agent Administration — GZ17-6.02 will be taken orally with a high-fat meal at a fixed dose of 375 mg twice daily each day of a 28-day cycle, continuing until progression or intolerable toxicity

SUMMARY:
The purpose of this clinical trial is to determine if GZ17-6.02 delays progression of castration-resistant prostate cancer.

DETAILED DESCRIPTION:
This single-arm phase Ib study will assess whether GZ17-6.02, a combination of curcumin, harmine, and isovanillin, delays radiographic progression of castration-resistant prostate cancer among men previously treated with androgen deprivation therapy and an androgen receptor pathway inhibitor. All participants in the study will receive GZ17-6.02. The study will also assess the safety and tolerability of GZ17-6.02 and explore patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with prostate cancer and treated with androgen deprivation therapy (ADT) and at least one androgen receptor pathway inhibitor (ARPI) (eg, abiraterone, enzalutamide, apalutamide or darolutamide). Previous prostate-specific membrane antigen (PSMA)-targeted therapy or cytotoxic chemotherapy is allowed but not required.
* Androgen levels ≤50 ng/dL (≤1.73 nmol/L).
* Disease progression following ADT and ARPI treatment described
* PSA progression over 2 assessments, defined as rising PSA values from 2 consecutive assessments with an interval of at least 7 days between assessments. PSA levels prior to study enrollment are considered and appropriate for inclusion.
* Measurable disease by RECIST v1.1 on chest/abdomen/pelvis CT or evaluable disease observed on bone scan.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Appropriate hepatic function defined by a total bilirubin (TBL) ≤1.5 × the upper limit of normal (ULN), alanine aminotransferase (ALT) AND aspartate aminotransferase (AST) ≤3 × ULN at screening.
* Appropriate kidney function defined by calculated or actual creatinine clearance ≥30 mL/min
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3.
* Platelets ≥100,000 cells/mm3.
* Serum hemoglobin level ≥8 g/dL.
* Agree to not donate blood or sperm during the study and for 90 days after the last dose of study treatment.
* Patients with sexual partners of childbearing potential must agree to use highly effective methods of contraception throughout the study
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Any investigational agent:

within 4 weeks OR within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, before initiating study treatment.

* Low PSA (≤10 ng/mL) at initial presentation (before ADT or at symptomatic progression in the castrate setting) plus high volume (≥20) bone metastases.
* Simultaneous enrollment in any other cancer treatment interventional clinical trial.
* Active, uncontrolled diarrhea leading to dehydration or electrolyte disturbances not controlled with oral repletion.
* Grade ≥3 uncontrolled infection.
* Major surgery (in the opinion of the treating investigator) ≤3 weeks before initiating study treatment.
* Not having fully recovered to a grade of 1 or lower from any surgery-related adverse effects within the 3 weeks preceding the start of the study treatment.
* Small cell, anaplastic, or neuroendocrine component.
* Known active brain metastasis.
* Known active leptomeningeal disease.
* Planned ongoing treatment with other drugs thought to potentially have adverse interactions with either of the medications included in the study treatment must be discontinued ≥2 weeks prior to initiating study treatment unless otherwise noted:

  * Monoamine oxidase inhibitors (MAOI) use; must discontinue use 10 days prior to initiating study therapy.
  * Strong or moderate CYP1A2, CYP3A4 and CYP2C19 inhibitors.
  * Rucaparib, Olaparib and Talazoparib, due to their common findings of liver enzyme elevation.
* Inability to swallow medication.
* Known hypersensitivity to GZ17-6.02 components (curcumin, harmine, and isovanillin) or excipients.
* Known or suspected malabsorption condition or obstruction.
* Active untreated hepatitis B or C" and "Known liver cirrhosis of any cause, active nonalcoholic steatohepatitis, or nonalcoholic fatty liver disease. Note: no additional testing necessary to confirm
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
Radiologic progression-free survival (rPFS) for 6 months or longer | 6 months and up to 5 years after end of study treatment
  Number of participants with rPFS for 6 months or longer

SECONDARY OUTCOMES:
Measure the biochemical response rate of CRPC tumors to GZ17-6.02 | Up to 5 years following end of study treatment
  Biochemical response measured by percentage of patients with any reduction in PSA, reduction in PSA by at least 30% (PSA30), and reduction in PSA by at least 50% (PSA50).
Measure the duration of response of CRPC tumors to GZ17-6.02 | Up to 5 years following end of study treatment
  Duration of tumor response, measured by time to increase in PSA.
Assess the objective response rate (ORR) in CRPC patients treated with twice daily GZ17-6.02. | Up to 5 years following end of study treatment
  Best objective response (complete response, partial response, or stable disease ≥4 months) in patients with measurable disease by RECIST 1.1.
Measure the duration of radiographic response in CRPC patients treated with twice daily GZ17-6.02 | Up to 5 years following end of study treatment
  Duration of radiographic response
Measure overall survival (OS) in CRPC patients treated with twice daily GZ17-6.02 | Up to 5 years following end of study treatment
  Overall patient survival, defined as date of diagnosis to date of death
Determine the safety and tolerability of twice daily treatment with GZ17-6.02 | Beginning of study treatment through the 30-day follow-up safety assessment up to 5 years
  Incidence of adverse events using Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: John Melson, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Currently, there are no plans to share IPD.